CLINICAL TRIAL: NCT05450601
Title: A Multicenter, Randomized, Doube-blind, Phase III Study to Evaluate the Efficacy and Safety of HCP2102 in Patients With Essential Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of HCP2102 in Essential Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALCH-302
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): HCP2102
  Interventions: Drug: HCP2102-1; Drug: HPP2104-1; Drug: HCP2102-2; Drug: HPP2104-2
- Active Comparator (Active Comparator): RLD2106
  Interventions: Drug: RLD2106-1; Drug: HPP2103-1; Drug: RLD2106-2; Drug: HPP2103-2

INTERVENTIONS:
Drug: HCP2102-1 — Take once daily for 2 weeks orally
  Arms: Experimental
Drug: HPP2104-1 — Placebo drug. Take once daily for 2 weeks orally
  Arms: Experimental
Drug: HCP2102-2 — Take once daily for 6 weeks orally
  Arms: Experimental
Drug: HPP2104-2 — Placebo drug. Take once daily for 6 weeks orally
  Arms: Experimental
Drug: RLD2106-1 — Take once daily for 2 weeks orally
  Arms: Active Comparator
Drug: HPP2103-1 — Placebo drug. Take once daily for 2 weeks orally
  Arms: Active Comparator
Drug: RLD2106-2 — Take once daily for 6 weeks orally
  Arms: Active Comparator
Drug: HPP2103-2 — Placebo drug. Take once daily for 6 weeks orally
  Arms: Active Comparator

SUMMARY:
A multicenter, randomized, double-blind, phase III study to evaluate the efficacy and safety of HCP2102 in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 19 years
2. Patients who understands the process of clinical study and voluntarily signs a peer letter
3. Visit 1: A person whose blood pressure measured in visit 1 corresponds to the following conditions

   * Blood pressure medication taken patients: 140mmHg ≤ sitSBP<200mmHg, sitDBP<120mmHg
   * Blood pressure medication free patients: 160mmHg ≤ sitSBP<200mmHg, sitDBP<120mmHg
4. Visit 2: 140mmHg ≤ sitSBP<200mmHg, sitDBP<120mmHg

Exclusion Criteria:

1. Difference between arms greater than 20 mmHg for mean sitSBP or 10 mmHg for mean sitDBP
2. Orthostatic hypotension with symptoms within 3 months prior to visit 1
3. Secondary hypertension patient or suspected to be
4. Uncontrolled diabetes mellitus(HbA1c > 9%) or type I diabetes mellitus
5. Active gout or hyperuricemia (uric acid ≥ 9mg/dL)
6. Severe heart disease or severe neurovascular disease
7. Severe or malignant retinopathy
8. Clinically significant hematological finding
9. Severe renal diseases (eGFR<30mL/min/1.73m2)
10. Severe hepatopathy or active hepatopathy (AST or ALT normal range ≥ 3 times)
11. Hypokalemia or Hyperkalemia(K<3.5mmol/L or K ≥ 5.5mmol/L)
12. Hyponatremia or Hypernatremia(Na<135mmol/L or Na ≥ 155mmol/L)
13. Hypercalcemia(Ca ≥ 10.5mg/dL)
14. History of malignancy tumor
15. History of autoimmune disease
16. History of alcohol or drug abuse
17. Positive to pregnancy test, nursing mother, intention on pregnancy
18. Considered by investigator as not appropriate to participate in the clinical study with other reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | week 8

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | week 2
Change from baseline in mean sitting diastolic blood pressure(mmHg) | week 2, 8
Change from baseline in mean pulse blood pressure(mmHg) | week 2, 8
Target blood pressure reaching rate(%) | week 2, 8
Blood pressure responder rate(%) | week 2, 8

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea